CLINICAL TRIAL: NCT07219017
Title: Mass Balance Study of [14C] ABBV-1354 (Icalcaprant) in Healthy Male Subjects Following Single Oral Dose Administration
Brief Title: A Study to Assess the Mass Balance of Oral ABBV-1354 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M25-571
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-1354

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-1354 (Experimental): Participants will receive a single dose of oral ABBV-1354 and followed 30 days post dose.
  Interventions: Drug: ABBV-1354

INTERVENTIONS:
Drug: ABBV-1354 — Oral solution

SUMMARY:
This study is to assess the mass balance of oral ABBV-1354 in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Male participants are eligible to participate if they agree to the following from Study Day 1 and for at least 93 days after the last dose of study treatment:
* Refrain from donating sperm

PLUS, either:

- Practice true abstinence, defined as: Refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable.

OR

* Use a male condom with spermicide (even with a successful vasectomy) with female partner who also uses a highly effective contraceptive method with a failure rate of < 1% per year (when used consistently and correctly).

AND

* Advise of the benefit for a female partner to use a highly effective method of contraception (as a condom may break or leak) if having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* BMI is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenths decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History: of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection, etc.].

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 32 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change from Baseline in Vital Sign Measurements | Up to approximately 15 days
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change From Baseline in Electrocardiograms (ECGs) | Up to approximately 15 days
  12-lead resting ECG will be recorded.
Number of Participants with Abnormal Change in Physical Examinations | Up to approximately 15 days
  Number of participants with abnormal change in physical examinations in areas like cardiovascular, respiratory, gastrointestinal, and neurological systems will be assessed.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to approximately 15 days
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Maximum observed concentration (Cmax) of ABBV-1354 | Up to approximately 15 days
  Cmax of ABBV-1354 will be assessed.
Time to Cmax (peak time, Tmax) of ABBV-1354 | Up to approximately 15 days
  Max of ABBV-1354 will be assessed.
Terminal phase elimination half-life (t1/2) of ABBV-1354 | Up to approximately 15 days
  Terminal phase elimination half-life (t1/2) of ABBV-1354 will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt) of ABBV-1354 | Up to approximately 15 days
  AUCt of ABBV-1354 will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to infinite time (AUCinf) of ABBV-1354 | Up to approximately 15 days
  AUCinf of ABBV-1354 will be assessed.
Amount of ABBV-1354 excreted in the urine over the sampling period (Aeu) | Up to approximately 15 days
  Amount of ABBV-1354 excreted in the urine over the sampling period (Aeu) will be assessed.
Percent of ABBV-1354 excreted in the urine | Up to approximately 15 days
  Percent excreted = 100 × (Aeu/dose).
Amount of ABBV-1354 excreted in the feces over the sampling period (Aeu) | Up to approximately 15 days
  Amount of ABBV-1354 excreted in the feces over the sampling period (Aeu) will be assessed.
Percent of ABBV-1354 radioactivity excreted in the feces | Up to approximately 15 days
  Percent excreted = 100 × (Aeu/dose).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Fortrea Clinical Research Unit Inc /ID# 277011, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-571